CLINICAL TRIAL: NCT00544349
Title: Phase II Study Evaluating the Effectiveness of the Association of Chemotherapy LV5FU2 Simplified and Cetuximab With Intra-arterial Hepatic Chemotherapy Using Oxaliplatin in Patients With Colorectal Cancer and Nonresectable Hepatic Metastases
Brief Title: Leucovorin, Fluorouracil, Cetuximab, and Oxaliplatin in Treating Patients With Stage IV Colorectal Cancer and Liver Metastases That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564063; FRE-IGR-CHOICE; IGR-1207; INCA-RECF0449
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; recurrent colon cancer; stage IV rectal cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as leucovorin, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving more than one drug (combination chemotherapy) and giving them together with cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving leucovorin together with fluorouracil, cetuximab, and oxaliplatin works in treating patients with stage IV colorectal cancer and liver metastases that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of this regimen by the measurement of objective response rate (RECIST criteria).

Secondary

* Determine the toxicity of this regimen.
* Evaluate the duration of tumor response.
* Determine the duration and rate of tumor control.
* Determine the rate of secondary resectability of hepatic metastases.
* Evaluate progression-free survival
* Determine rate of progression of the tumor.
* Determine overall survival.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1 hour, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours. Patients also receive oxaliplatin by hepatic arterial infusion over 2 hours. Treatment continues for at least 3 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary cancer of the colon or rectum

  * Isolated hepatic metastases
  * Not amenable to curative resection or requirement for complex and or larger (i.e., > 4 liver segments) liver resection
* Measurable disease (RECIST criteria)
* Original tumor must be (or have been) removed

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-1
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 times normal
* Bilirubin ≤ 1.5 times upper limit of normal
* Transaminases ≤ 5 times normal
* Not pregnant or nursing
* Fertile patients must use effective contraception

Exclusion criteria:

* Contraindication or allergy grade 3-4 to any components of the study drugs
* Peripheral neuropathy
* Intestinal occlusion or subocclusion or prior inflammatory intestinal disease
* Severe cardiac disease including any of the following:

  * Symptomatic coronary disease
  * Myocardial infarction in the past 6 months
  * New York Heart Association grade II-IV cardiac insufficiency
  * Severe arrhythmia (even if treated)
* Active or uncontrolled infection
* Other concurrent serious disorder
* Severe uncontrolled medical condition
* Other malignancy within the past 5 years or concurrently except basal cell skin cancer or carcinoma in situ of the cervix
* Study impossible due to psychological, geographical, or social reasons
* Prisoners or patients under guardianship

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Prior chemotherapy except adjuvant chemotherapy comprising fluorouracil, leucovorin calcium, capecitabine, oxaliplatin, irinotecan hydrochloride, and/or bevacizumab (completed > 6 months ago if oxaliplatin- or irinotecan-based)
* Prior epidermal growth factor (EGF), monoclonal antibody inhibiting transduction of EGF receptor (EGFR), or any other treatment targeting the EGFR
* Other concurrent anticancer immunotherapy, chemotherapy, or hormone therapy
* Participation in another study in the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: objective tumor response rate (RECIST criteria)

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0
Duration of response
Duration and rate of tumor control
Secondary resectability of hepatic metastases
Progression-free survival
Overall survival
Tumor progression rate

CONTACTS AND LOCATIONS:
Overall Officials: David Malka, MD, PhD — Gustave Roussy, Cancer Campus, Grand Paris
Locations (7):
- France (7):
  - Hopital Saint Andre, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - CHU Pitie-Salpetriere, Paris
  - Centre Eugene Marquis, Rennes
  - Hopital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif